CLINICAL TRIAL: NCT02381977
Title: Prevalence of Acute Critical Neurological Disease in Children: a Global Epidemiological Assessment
Acronym: PANGEA
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Principal Investigator, Ericka Fink, Associate Professor, Pediatric Critical Care Medicine, University of Pittsburgh
Other Study IDs: PANGEA
Record Dates: First submitted 2015-02-16; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Cardiac Arrest; Stroke; Traumatic Brain Injury; Brain Mass; Status Epilepticus; Spinal Cord Disease; Hydrocephalus
MeSH Terms: conditions — Heart Arrest; Stroke; Brain Injuries, Traumatic; Status Epilepticus; Spinal Cord Diseases; Hydrocephalus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
PANGEA is an international prospective point prevalence study to describe the epidemiology, interventions, and outcomes in children with acute critical brain disease.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7 days to 17 years inclusively and admitted to an ICU (ICU can be classified as general, cardiac, trauma, etc).
2. Children with acute or acute on chronic neurologic disease that occurred just prior to hospital admission or occurred during the hospital admission.
3. Acute neurologic disease is secondary to TBI, stroke, brain mass, hydrocephalus, cardiac arrest, status epilepticus, CNS infection/inflammation, or spinal cord injury.

Exclusion Criteria:

1. Children with acute perinatal neurologic disease.
2. Children with isolated chronic brain injury and no acute neurologic disease.

Ages: 7 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically-ill children with acute neurologic injury
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of acute brain insult | 4 days over a 1 year period

SECONDARY OUTCOMES:
Mortality | Hospital discharge or 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ericka Fink, MD, MS, Principal Investigator — 4126925164